CLINICAL TRIAL: NCT03936049
Title: Replication of the LEADER Diabetes Trial in Healthcare Claims
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-LEADER
Record Dates: First submitted 2019-04-29; First posted 2019-05-03 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Liraglutide; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DPP-4 inhibitor: Reference group
  Interventions: Drug: DPP-4 inhibitor
- Liraglutide: Exposure group
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Liraglutide dispensing claim is used as the exposure group
  Groups: Liraglutide
Drug: DPP-4 inhibitor — DPP-4 inhibitor dispensing claim is used as the reference group
  Groups: DPP-4 inhibitor

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see: https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Eligible cohort entry dates Market availability of liraglutide in the U.S. started on January 20, 2010. For Marketscan and Medicare: January 20, 2010-Dec 31, 2016 (end of data availability).

For Optum: January 20, 2010-Sep 30, 2017 (end of data availability).

Inclusion Criteria:

* Men or women with type 2 diabetes
* Either of the following:

  * Prior cardiovascular disease cohort: Age ≥ 50 years at screening, AND at least one of the following:

    * Prior MI
    * Prior stroke or TIA
    * Prior coronary, carotid or peripheral arterial revascularization
  * >50% stenosis of coronary, carotid, or lower extremity arteries coded by Peripheral vascular disease
  * Chronic heart failure NYHA class II-III
  * CKD stage 3-6 as Chronic renal failure:
* No Prior cardiovascular disease group: Age ≥ 60 years at screening, AND at least one of the following:

  * Microalbuminuria or proteinuria
  * Hypertension and left ventricular hypertrophy by ECG or imaging
  * Ankle-brachial index <0.9

Exclusion Criteria:

* Type 1 diabetes
* Use of a GLP-1 receptor agonist (exenatide, liraglutide or other) or pramlintide or any (dipeptidyl peptidase 4 (DPP-4) inhibitor within the 3 months prior to screening
* Use of long-term insulin in 90 days prior
* Diabetic ketoacidosis in 3 months prior to index date as Acute decompensation of glycaemic control requiring immediate intensification of treatment to prevent acute complications of diabetes (e.g., diabetic ketoacidosis) in the previous 3 months
* Inpatient (hospitalization) code for MI, stroke, revascularization, PTCA, CABG IN PRIOR 14 DAYS as An acute coronary or cerebrovascular event in the previous 14 days
* inpatient Heart failure (CHF) as Chronic heart failure NYHA class IV
* ESRD codes as Current continuous renal replacement therapy
* Liver disease as "End stage liver disease, defined as the presence of acute or chronic liver disease and recent history of one or more of the following: ascites, encephalopathy, variceal bleeding, bilirubin ≥ 2.0 mg/dL, albumin level ≤ 3.5 g/dL, prothrombin time ≥ 4 seconds prolonged, international normalised ratio (INR) ≥1.7 or prior liver transplant"
* Organ transplant codes as A prior solid organ transplant or awaiting solid organ transplant
* History of malignant neoplasm in previous 5 years 140.xx-208.xx (except 173.xx, non-melanoma skin cancer)
* Family or personal history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma (FMTC)
* Personal history of non-familial medullary thyroid carcinoma
* Drug abuse or dependence as Known use of non prescribed narcotics or illicit drugs
* Encounter for contraceptive management, Oral contraceptives, and pregnancy as "Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures as required by local law or practice)"

Ages: 50 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, cohort study design comparing liraglutide to the DPP4 inhibitor (DPP4i) antidiabetic class as a proxy for placebo. Both 2nd generation sulfonylureas (SUs) and DPP4is are not known to have an impact on the outcome of interest. The comparison against DPP4i is the primary comparison. Initiators of 2nd generation SUs are used as a secondary comparator group. The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of liraglutide or a comparator drug (cohort entry date). Follow-up for the outcome (3P-MACE), begins the day after drug initiation. As in the trial, patients are allowed to take other antidiabetic medications during the study.
Sampling Method: Non-Probability Sample
Enrollment: 168690 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Relative hazard of composite outcome of Stroke, MI, and Mortality | Through study completion (a median of 154-188 days)
  Relative hazard of composite outcome of MI, stroke, and mortality - Please refer to uploaded protocol for full definition due to size limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham And Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Franklin JM, Patorno E, Desai RJ, Glynn RJ, Martin D, Quinto K, Pawar A, Bessette LG, Lee H, Garry EM, Gautam N, Schneeweiss S. Emulating Randomized Clinical Trials With Nonrandomized Real-World Evidence Studies: First Results From the RCT DUPLICATE Initiative. Circulation. 2021 Mar 9;143(10):1002-1013. doi: 10.1161/CIRCULATIONAHA.120.051718. Epub 2020 Dec 17. PMID 33327727

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT03936049/Prot_SAP_003.pdf